CLINICAL TRIAL: NCT03634644
Title: Omega-3 Polyunsaturated Fatty Acids for the Treatment of Patients With Idiopathic Oligoasthenoteratospermia: A Double-blind, Placebo-controlled and Randomized Exploratory Clinical Trial
Brief Title: Omega-3 PUFA for Treatment of Patients With Idiopathic Oligoasthenoteratospermia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Bing Yao, Director of Center for Reproductive Medicine, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Omeag-3PUFA for OAT
Record Dates: First submitted 2018-08-12; First posted 2018-08-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Male Infertility Due to Hypospermatogenesis
Keywords: male infertility; oligoasthenoteratospermia
MeSH Terms: conditions — Infertility, Male | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acid capsule (Active Comparator): 1g per capsule(EPA400mg，DHA320mg)
  Interventions: Drug: Omega 3 fatty acid
- Placebo capsule (Placebo Comparator): The placebo capsule has same appearance and packing with the Omega-3 fatty acid capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Omega 3 fatty acid — Omega 3 fatty acid,mainly composed of EPA and DHA.
  Other Names: Placebo Capsule
  Arms: Omega-3 fatty acid capsule
Drug: Placebo oral capsule — mainly composed of corn oil
  Arms: Placebo capsule

SUMMARY:
Investigators have previously found that sperm quality was not related to obesity indicators, such as body mass index (bmi), waist circumference, waist-hip ratio, girth ratio and serum lipid, but seminal plasma lipids could notably affect the sperm concentration, sperm progressive ratio(PR), sperm DNA fragmentation index (DFI). These results indicates that abnormal lipid metabolism in the male reproductive system may affect male fertility.

It seems that the sperm fatty acid spectrum is associated with n-3 polyunsaturated fatty acids (PUFA) in dietary. Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA) are the most common n-3 PUFA. Only plasma DHA/EPA may reflect the quantity of DHA/EPA in adults. Most research indicate that n-3 PUFA is the main polyunsaturated fatty acid in human sperm.

It is well known that diets have great influence on the gut microbiota composition. Many researches have delineated the cause and effect relationship between disturbed gut microbes and diseases, such as irritable bowel syndrome, obesity, diabetes. The disturbed gut microbiota ecosystem may also lead to the intestinal mucosal permeability increasing, which may result in endotoxemia and a series of metabolic syndrome. N-3 polyunsaturated fatty acids may play an important role in regulating metabolism and physiological functions in the body. A clinical research found that both total n-3 PUFA and DHA serum levels were significantly correlated with microbiome alpha diversity. Therefore, investigators may try to figure out the influence of n-3 PUFA supplement on gut microbiota composition and whether the gut microbiota have influence on sperm parameters. So investigators apply for your permission to collected the fecal samples from the participants, which will be a meaningful work.

DETAILED DESCRIPTION:
In the previous work, investigators found high fat diet induced gut microbiota dysbiosis can lead to low sperm motility and sperm count, and also recognised some microbes which may lead to the low sperm motility and sperm count. It is obvious that gut microbiota can influence the sperm quality. And the supplement of n-3 PUFA is significantly correlated with microbiome alpha diversity. So investigators want to collected the fecal samples from the participants, to ascertain whether the supplementation of n-3 PUFA can promote sperm parameters by improve gut microbiota ecosystem.

The potential microbes planing to cultivate: Prevotella spp, bacteroides spp.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Oligoasthenoteratospermia.

Exclusion Criteria:

* Leukocytospermia, prostatitis, genital trauma, testicular torsion, urinary tract infections, cryptorchidism, varicocele, diabetes, inguinal and genital surgery.
* Y chromosome microdeletion and chromosomal karyotype abnormality.
* Extreme oligospermia.
* Hepatobiliary diseases, kidney failure.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2022-10-28 (Estimated)

PRIMARY OUTCOMES:
sperm concentration | 40 days
  sperm concentration

SECONDARY OUTCOMES:
progressive ratio | 40 days
  progressive sperm concentration/total sperm concentration

OTHER OUTCOMES:
DNA fragmentation index | 40 days
  DNA fragmentation index
gut microbiota composition | 40 days
  variation of gut microbiota composition collecting from patients' fecal sample

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Reproductive Medicine, Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ding N, Zhang X, Zhang XD, Jing J, Liu SS, Mu YP, Peng LL, Yan YJ, Xiao GM, Bi XY, Chen H, Li FH, Yao B, Zhao AZ. Impairment of spermatogenesis and sperm motility by the high-fat diet-induced dysbiosis of gut microbes. Gut. 2020 Sep;69(9):1608-1619. doi: 10.1136/gutjnl-2019-319127. Epub 2020 Jan 2. PMID 31900292